CLINICAL TRIAL: NCT02365558
Title: Evaluation of the Impact of Increased Gastric pH Following Omeprazole Administration on the Pharmacokinetics of Evacetrapib in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of Increased Stomach pH on Evacetrapib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15373; I1V-MC-EIBO (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-02-06; First posted 2015-02-19 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-02

CONDITIONS: Healthy
MeSH Terms: interventions — evacetrapib; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evacetrapib (Experimental): Single oral dose of evacetrapib administered alone on Day 1 of Period 1.
  Interventions: Drug: Evacetrapib
- Omeprazole + Evacetrapib (Experimental): In Period 2, participants will receive 40 mg oral dose of Omeprazole once daily (QD) on Days 8 through 20.
  Evacetrapib will be co-administered once, orally on Day 14.
  Interventions: Drug: Evacetrapib; Drug: Omeprazole

INTERVENTIONS:
Drug: Evacetrapib — Administered orally
  Other Names: LY2484595
Drug: Omeprazole — Administered orally
  Arms: Omeprazole + Evacetrapib

SUMMARY:
The purpose of this study is to evaluate the effect of increased stomach pH on how much evacetrapib is found in the blood stream and how long the body takes to get rid of it when given to healthy participants. Information about any side effects that may occur will also be collected.

There are two parts to the study. Participation in both parts will be required.

The study will last approximately 30 days, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy participants, as determined by medical history and physical examination
* Females must be of non-child-bearing potential
* Have a body mass index of 18 to 32 kilograms per square meter (kg/m^2)

Exclusion Criteria:

* Have known allergies to evacetrapib, omeprazole, related compounds, or any components of the evacetrapib or omeprazole formulations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Evacetrapib: Evacetrapib 130 milligram (mg) administered as a single oral dose on Day 1.
- Evacetrapib + Omeprazole: Omeprazole 40 mg administered once daily (QD) orally on Day 8 through 20. Evacetrapib 130mg coadministered as a single oral dose on Day 14.
Period: Period 1 (Day 1 Through Day 7)
Arm/Group | Evacetrapib | Evacetrapib + Omeprazole
Started | 34 | 0
Received at Least One Dose of Study Drug | 34 | 0
Completed | 33 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2 (Day 8 Through Day 20)
Arm/Group | Evacetrapib | Evacetrapib + Omeprazole
Started | 0 (Participants move to Evacetrapib + Omeprazole for Period 2.) | 33 (Participants completed Period 1 and entered Evacetrapib + Omeprazole for Period 2.)
Completed | 0 | 32
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Single oral dose of 130 mg evacetrapib on Day 1 and oral doses of 40 mg omeprazole QD on Days 8 through 20, with a single oral dose of 130 mg evacetrapib coadministered on Day 14
Arm/Group | Overall Study
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Evacetrapib
Time Frame: Day 1 and Day 14 at 0, 1, 2, 3, 4, 6, 8,12, 24, 36, 48, 72, 96, 120, 144 and 168 Hours Postdose
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Evacetrapib: Single oral dose of Evacetrapib administered on Day 1 of Period 1
- Evacetrapib + Omeprazole: In Period 2, Participants will receive 40 mg oral dose of Omeprazole QD on Days 8 through 20.
  Evacetrapib will be coadministered once, orally on Day 14.
Arm/Group | Evacetrapib | Evacetrapib + Omeprazole
Number analyzed (Participants) | 34 | 33
nanograms per milliliter (ng/mL) | 748 (79) | 959 (88)

2. Primary Outcome: Pharmacokinetics (PK): Time of Maximum Observed Concentration (Tmax) of Evacetrapib
Time Frame: Day 1 and Day 14 at 0, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 Hours Postdose
Population: All participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: Hours
Groups:
- Evacetrapib + Omeprazole: In Period 2, participants will receive 40 mg oral dose of Omeprazole once daily (QD) on Days 8 through 20.
  Evacetrapib will be co-administered once, orally on Day 14.
Arm/Group | Evacetrapib | Evacetrapib + Omeprazole
Number analyzed (Participants) | 34 | 33
Hours | 3.00 [2.00 to 6.00] | 3.00 [1.00 to 6.00]

3. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞])
Time Frame: Day 1 and Day 14 at 0, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 and 168 Hours Postdose
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng·h/mL)
Arm/Group | Evacetrapib | Evacetrapib + Omeprazole
Number analyzed (Participants) | 34 | 33
nanogram*hour per milliliter (ng·h/mL) | 12400 (52) | 14100 (66)

ADVERSE EVENTS:
Groups:
- Evacetrapib + Omeprazole: In Period 2, participants will receive 40 mg oral dose of Omeprazole once daily (QD) on Days 8 through 20.
  Evacetrapib will be coadministered once, orally on Day 14.
  Evacetrapib: Administered orally
  Omeprazole: Administered orally
- Evacetrapib + Omeprazole Follow-up: Evacetrapib + Omeprazole Follow-up will occur at least 14 days after last dose of Evacetrapib on Day 14.
Arm/Group | Evacetrapib | Evacetrapib + Omeprazole | Evacetrapib + Omeprazole Follow-up
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 5/34 | 2/33 | 3/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evacetrapib (N=34) | Evacetrapib + Omeprazole (N=33) | Evacetrapib + Omeprazole Follow-up (N=33)
Vessel puncture site reaction (General disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No